CLINICAL TRIAL: NCT03440476
Title: Personalized Booster Feedback After Alcohol Health Education
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abby Braitman (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Abby Braitman, Assistant Professor, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-267; K01AA023849 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: College Student Drinking
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Masking Description: The intervention is an online program, not an individual, so masking is not necessary. Similarly, the same online survey is deployed in all follow-up assessments regardless of condition, and data are not collected by individuals, so masking is not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention-only Control (Placebo Comparator): Participants navigate through e-checkup to go, the well-established alcohol intervention. Their email 2 weeks later contains only a reminder to participate in follow-up surveys.
  Interventions: Behavioral: e-checkup to go
- Intervention plus feedback booster (Active Comparator): Participants navigate through e-checkup to go, the well-established alcohol intervention, then receives the Feedback-only booster. Their email 2 weeks later contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, their own use, and harm reduction strategies. The content is clearly automatically generated.
  Interventions: Behavioral: e-checkup to go; Behavioral: Feedback-only booster
- Intervention plus feedback and personal contact booster (Active Comparator): Participants navigate through e-checkup to go, the well-established alcohol intervention, then receives the Feedback-plus-personal-contact booster. Their email 2 weeks later contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, their own use, and harm reduction strategies. The email is sent from a member of the research staff.
  Interventions: Behavioral: e-checkup to go; Behavioral: Feedback-plus-personal-contact booster

INTERVENTIONS:
Behavioral: e-checkup to go — The e-checkup to go substance program is designed to motivate individuals to reduce their consumption using personalized information about their own use and risk factors. The program is a combination of several components including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It is self-guided and requires no face-to-face time with an administrator. It provides tailored feedback regarding quantity and frequency of alcohol use, normative comparisons, physical health information, amount and percent of income spent on alcohol, negative consequences feedback, explanation and advice for how to reach their goals, and resources.
Behavioral: Feedback-only booster — Booster emails will contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, their own reported consumption, and reminders of strategies they can use to protect themselves from alcohol-related harm. The content is clearly automatically generated.
  Arms: Intervention plus feedback booster
Behavioral: Feedback-plus-personal-contact booster — Booster emails will contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, their own reported consumption, and reminders of strategies they can use to protect themselves from alcohol-related harm. The email is sent from an individual on the research staff.
  Arms: Intervention plus feedback and personal contact booster

SUMMARY:
Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from heavy alcohol use can be mild (e.g., hangovers, missed classes), to severe (e.g., assault, even death). Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. Online interventions are cost-effective, offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment.

In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention (Braitman & Henson, 2016). Although promising, the booster incorporated in the study needs further empirical refinement.

The current project seeks to build on past progress by further developing and refining the booster. In particular, one aspect missing from online interventions is a connection with a person invested in improving the student's outcomes. The current study aims to generate a personal connection for online interventions through a follow-up booster emailed by a member of the research staff. Outcomes will be compared for participants who receive a follow-up booster with similar content, but is clearly automatically generated and not from any particular individual.

There are 3 conditions: all participants receive the initial online intervention targeting college drinking. Condition 1 (the control group) receives an email with a reminder to complete the follow-up surveys, but no feedback (i.e., no booster). Condition 2 receives an emailed booster with normative feedback plus protective strategies feedback, clearly automatically generated. Condition 3 receives an emailed booster with normative feedback plus protective strategies feedback, from a member of the research staff. The booster content alone (automatically generated) may be efficacious, or the additional personal connection may enhance the effect.

Thus, the aim of the current study is to examine if personal contact enhances the tailored feedback received via booster email.

DETAILED DESCRIPTION:
Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from frequent or heavy alcohol use can be mild (e.g., hangovers, missed classes), moderate (e.g., poor grades, damaged relationships), or severe (e.g., assault, even death). Given the potentially dangerous consequences, reducing alcohol use and associated problems is a major health priority. Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. The benefits of online interventions include cost-effectiveness and ease of administration, plus they offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment.

Although post-intervention boosters have been shown to be effective for individuals seeking treatment for alcohol-related injuries in emergency medical settings, limited studies have investigated the efficacy of boosters for college students who have received alcohol interventions. In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention, while at the same time maintaining low cost and easy dissemination (Braitman & Henson, 2016). Although promising, the booster incorporated in the study needs further empirical refinement.

The current project seeks to build on past progress reducing the gap between online and more efficacious in-person interventions. The current study further develops and refines the booster to identify optimal administration for maximum efficacy. In particular, one aspect missing from online interventions is a connection with a person invested in improving the student's outcomes. The current study aims to generate a personal connection for online interventions through a follow-up booster emailed by a member of the research staff. Outcomes will be compared for participants who receive a follow-up booster with similar content, but is clearly automatically generated and not from any particular individual.

There are 3 conditions: all participants receive the initial online intervention targeting college drinking. Condition 1 (the control group) receives an email with a reminder to complete the follow-up surveys, but no feedback (i.e., no booster). Condition 2 receives an emailed booster with normative feedback plus protective strategies feedback, clearly automatically generated. Condition 3 receives an emailed booster with normative feedback plus protective strategies feedback, from a member of the research staff. The booster content alone (automatically generated) may be efficacious, or the additional personal connection may enhance the effect.

Thus, the aim of the current study is to examine if personal contact enhances the tailored feedback received via booster email.

Hypothesis 1a: Both groups receiving emailed feedback will reduce drinking and alcohol-related problems as compared to the intervention-only control condition.

Hypothesis 1b: Reductions in drinking and problems will be stronger for those who receive emails from an individual rather than automatically generated.

ELIGIBILITY:
Inclusion Criteria:

* Current college students at the sponsor institution at the time of enrollment
* Between the ages of 18 and 24
* Consumed at least standard drink of alcohol in the past 2 weeks

Exclusion Criteria:

* Under age of 18
* Over age of 24
* Not a college student
* Did not drink alcohol in the past 2 weeks

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | Past 2 weeks
  Participant self-reported number of standard drinks consumed by participant over the past 2 weeks.

SECONDARY OUTCOMES:
Alcohol-related consequences | Past 2 weeks
  Participant self-report on the Young Adult Alcohol Consequences Questionnaire (YAACQ; Read, Kahler, Strong, & Colder, 2006), which assesses alcohol-related problems experienced by the participant. Total scores are created by summing all individual items, and range from 0 to 48, with higher values representing more problems experienced (i.e., worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Abby L Braitman, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03440476/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03440476/SAP_000.pdf
  • Informed Consent Form (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03440476/ICF_002.pdf